CLINICAL TRIAL: NCT02183896
Title: Efficacy of PRP (Platelet Rich Plasma) Following Arthroscopic Microfracture of Chondral Lesions of the Hip
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-0080
Record Dates: First submitted 2014-07-01; First posted 2014-07-08 (Estimated); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Femoroacetabular Impingement; Chondral Lesions
Keywords: Femoroacetabular impingement (FAI); Chondral lesions; Hip; Microfracture; Platelet-rich plasma (PRP)
MeSH Terms: conditions — Femoracetabular Impingement; Fractures, Stress | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- Platelet-rich plasma (PRP) (Experimental): Intra-articular injections in the hip of autologous platelet-rich plasma (PRP) at week 1 and 2 post-operatively. Dose 5 mL. PRP is derived from the patient's own blood.
  Interventions: Biological: Platelet-rich plasma (PRP)
- Saline (Placebo Comparator): Intra-articular injections in the hip of saline, solution week 1 and 2 post-operatively. Dose: 5 mL at each injection.
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: Platelet-rich plasma (PRP)
  Other Names: PRP; Autologous platelet-rich plasma; Autologous PRP
  Arms: Platelet-rich plasma (PRP)
Drug: Saline
  Other Names: 0.9% Sodium Chloride
  Arms: Saline

SUMMARY:
The purpose of this research project is to assess the effectiveness of intra-articular injections of autologous platelet-rich plasma (PRP) after arthroscopic microfracture. Our hypothesis is that platelet-rich plasma will improve patient's clinical outcomes and chondral healing following microfracture performed during femoroacetabular impingement (FAI) hip arthroscopy.

DETAILED DESCRIPTION:
The purpose of this research project is to assess the effectiveness of intra-articular injections of autologous platelet-rich plasma (PRP) after arthroscopic microfracture. Our hypothesis is that platelet-rich plasma will improve patient's clinical outcomes and chondral healing following microfracture performed during femoroacetabular impingement (FAI) hip arthroscopy.

This study has two aims:

1. Evaluate clinical efficacy of intra-articular injections of platelet-rich plasma (PRP) following arthroscopic microfracture.
2. Evaluate if microfracture followed by PRP injections improves chondral healing.

Microfracture has shown good results with chondral lesions of the hip. However, microfracture does not regenerate normal hyaline cartilage. There is growing evidence that PRP can improve articular cartilage healing. Injection of PRP following microfracture may help regeneration to normal hyaline like articular cartilage together with soft tissue healing, thereby improving patients' early and long-term outcomes of chondral healing.

Patients will be randomized to one of two study arms - microfracture with PRP (treatment arm) and microfracture with saline (control arm) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18-50, inclusive.
2. Healthy patients undergoing hip arthroscopy due to FAI.
3. No OA according to X-Ray, defined by the presence of joint space narrowing, osteophytes, sclerosis and subchondral cysts and surgery observation (Tonnis grade 0-1).
4. No other influential disabilities in lower limbs, which could alter the post-operative therapy.
5. No chronic use of NSAIDs, steroids, or chemotherapy drugs during the last 6 months before enrollment.
6. Women of childbearing potential will be allowed to enroll but must be willing to practice one highly effective method of contraception (oral, injectable or implanted hormonal methods of contraception, placement of an intrauterine device [IUD] or intrauterine system [IUS] condom or occlusive cap with spermicidal foam/gel/film/cream/suppository, male sterilization, or true abstinence) throughout the study.
7. Intra-articular cartilage lesion grade 2-3-4-5 of Beck Classification or III-IV of Outerbridge.

Exclusion Criteria:

1. Patients with autoimmune concomitant disease(s) that may affect joints, such as rheumatoid arthritis (RA), psoriatic arthritis and lupus arthritis.
2. Patients with polyarticular disease.
3. Patients with major conditions, such as poorly controlled diabetes, congestive heart failure (CHF), chronic obstructive pulmonary disease (COPD) or untreated depression.
4. Patients with blood disorders (thrombopathy, thrombocytopenia, anemia with hemoglobin <9g/dL).
5. Patients who had intra-articular treatment with steroids within 6 months of enrollment in this study or received more than 3 previous intra-articular steroid injections to the effected hip.
6. Patients who are pregnant or nursing at the time of consent.
7. Non-English speaking patients. (Scores used for evaluation have not been validated in Spanish).
8. Patients who had previous hip surgery.
9. Additional disabilities in any of the lower limbs that would interfere with any of the clinical assessments.
10. Chronic use of NSAIDs (defined as taking NSAID regularly every week for the last 6 months), steroids or chemotherapy drugs.
11. Patients with a BMI over 30. Due to the fact that this study utilizes an injection technique, which may be inaccurate in obese subjects.
12. Patients with pacemakers or metal implants who are unable to get an MRI.
13. Non-adherence according to inclusion criteria.
14. Patients allergic to lidocaine

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
MRI dGEMRIC | 12 and 24 months post-operative
  MRI dGEMRIC will be utilized to assess chondral healing. Change is being assessed between measurement time points.

SECONDARY OUTCOMES:
PA Hip X-Ray | Baseline, 12 and 24 months post-operative
  Change is being assessed between measurement time points.
International Hip Outcome Tool (IHOT) | Pre-operative; and 3, 6, 12, and 24 month post-operative
  Patient reported outcomes assessed from patient completed surveys. Change is being assessed between measurement time points.
Western Ontario and McMaster (WOMAC) osteoarthritis index | Pre-operative; and 3, 6, 12, and 24 month post-operative
  Patient reported outcomes assessed with patient completed survey.Change is being assessed between measurement time points.
Non-arthritic hip score | Pre-operative; and 3, 6, 12, and 24 month post-operative
  Patient reported outcomes assessed with patient completed survey. Change is being assessed between measurement time points.
Range of Motion (ROM) | Pre-operative; prior to injections at week 1 and 2 post-operative; 6 week, and 3, 6, 12, and 24 months post-operative
  ROM assessed as part of clinical outcome physical exam. Change is being assessed between measurement time points.
Flexion Abduction and External Rotation (FABER) | Pre-operative; prior to injections at week 1 and 2 post-operative; 6 week, and 3, 6, 12, and 24 months post-operative
  FABER assessed as part of clinical outcome physical exam. Change is being assessed between measurement time points.
Bicycle Kicks | Pre-operative; prior to injections at week 1 and 2 post-operative; 6 week, and 3, 6, 12, and 24 months post-operative
  Bicycle kicks assessed as part of clinical outcome physical exam. Change is being assessed between measurement time points.

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Pascual-Garrido, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, CU Sports Medicine, Boulder, Colorado, United States